CLINICAL TRIAL: NCT02244359
Title: Improving the Decision Making Process About Location of Care With the Frail Elderly and Their Caregivers
Brief Title: Improving Decision Making On Location of Care With the Frail Elderly and Their Caregivers
Acronym: DOLCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: TVN 2013 Core Research Grant Program (Unknown); Ministere de la Sante et des Services Sociaux (Other); Health and Social Services Agency, Montreal (Other)
Responsible Party: Principal Investigator, France Legare, B. Sc. Arch, MD, PhD, CCMF, FCMF, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CORE 2013-56
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Decision Process About the Location of Care Among Frail Elderly
Keywords: Shared Decision making; Patient Centred care; Interprofessionalism; Home care; Frail elderly

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Training (Experimental): Online tutorial, decision aid and interactive workshop
  Interventions: Behavioral: Training
- Usual care (Other): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Training
  Arms: Training
Behavioral: Usual care
  Arms: Usual care

SUMMARY:
One of the toughest decisions faced by the frail elderly in Canada is whether to stay at home or move to a care facility. It is certainly difficult to make this decision alone, but can be even harder if someone else makes it for you. Shared decision making is when, instead of making decisions for the patient, healthcare professionals share information about what the evidence says, and they talk about what's important with the patient, and then make the decision together. In the case of the frail elderly in home care services, there are many health care professionals involved, e.g. the doctor, nurse and social worker. In this case decisions should be shared by all the professionals involved with the elderly person along with his or her caregivers. Unfortunately, in this context, shared decision making rarely occurs.

We have designed a training program that teaches interprofessional teams how to share decisions with their frail elderly patients, and tested it in one Quebec City and one Edmonton home care team. This project tests the training program on a broader scale with 16 home care teams attached to community health centres across the province of Quebec, and will compare the results with what happens when no one has completed the training (usual care). Home care is a rapidly growing sector and this study will lay the foundations for a national strategy to ensure that no one has to make this difficult decision alone.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care from the home care team
* Faced the decision about whether to stay at home or move to a care facility in the previous 3 to 6 months
* Able to read, understand and write french or english
* Able to give informed consent
* For the case of clients unable to provide informed consent, their caregivers who was involved into decision making process will be eligible

Exclusion Criteria:

* Clients who cannot provide informed consent (e. g. clients with cognitive impairment) without a caregiver
* Clients who require acute care hospitalization and whom the location of care decision is transferred to hospital-based social services

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 455 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The assumed role in the decision making process, and the preferred and chosen options. | 3 to 6 months
  We will use the modified version of the Control Preferences Scale designed to assess the assumed role in the decision making process reported by the client.

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, MD, PhD, Principal Investigator — CHUQ Research Center
Locations (1):
- CHU de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Adekpedjou R, Haesebaert J, Stacey D, Briere N, Freitas A, Rivest LP, Legare F. Variations in factors associated with healthcare providers' intention to engage in interprofessional shared decision making in home care: results of two cross-sectional surveys. BMC Health Serv Res. 2020 Mar 12;20(1):203. doi: 10.1186/s12913-020-5064-3. PMID 32164669
- [Derived] Boucher A, Haesebaert J, Freitas A, Adekpedjou R, Landry M, Bourassa H, Stacey D, Croteau J, Genevieve PG, Legare F. Time to move? Factors associated with burden of care among informal caregivers of cognitively impaired older people facing housing decisions: secondary analysis of a cluster randomized trial. BMC Geriatr. 2019 Sep 9;19(1):249. doi: 10.1186/s12877-019-1249-1. PMID 31500590
- [Derived] Garvelink MM, Emond J, Menear M, Briere N, Freitas A, Boland L, Perez MMB, Blair L, Stacey D, Legare F. Development of a decision guide to support the elderly in decision making about location of care: an iterative, user-centered design. Res Involv Engagem. 2016 Jul 19;2:26. doi: 10.1186/s40900-016-0040-0. eCollection 2016. PMID 29062524
- [Derived] Garvelink MM, Freitas A, Menear M, Briere N, Stacey D, Legare F. In for a penny, in for a pound: the effect of pre-engaging healthcare organizations on their subsequent participation in trials. BMC Res Notes. 2015 Dec 8;8:751. doi: 10.1186/s13104-015-1743-2. PMID 26645477
- [Derived] Legare F, Briere N, Stacey D, Bourassa H, Desroches S, Dumont S, Fraser K, Freitas A, Rivest LP, Roy L. Improving Decision making On Location of Care with the frail Elderly and their caregivers (the DOLCE study): study protocol for a cluster randomized controlled trial. Trials. 2015 Feb 12;16:50. doi: 10.1186/s13063-015-0567-7. PMID 25881122